CLINICAL TRIAL: NCT02439905
Title: The Effects of Dexmedetomidine on Inflammatory Mediators After One Lung Ventilation During Video-assisted Thoracoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201410035MINC
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: One Lung Ventilation in Thoracic Surgery
Keywords: inflammatory cytokine; protective effect; Dexmedetomidine; Precedex; one lung ventilation; ischemia-reperfusion
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidine
- Normal saline group (Placebo Comparator)
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: Dexmedetomidine — In dexmedetomidine group, dexmedetomidine infusion starts at the time after induction of general anesthesia and before one lung ventilation. The infusion has continued until end of the operation.
  Arms: Dexmedetomidine group
Drug: Placebo control — In normal saline group, normal saline infusion starts at the time after induction of general anesthesia and before one lung ventilation. The infusion has continued until end of the operation.
  Arms: Normal saline group

SUMMARY:
During lung surgery, mechanical one-lung ventilation is usually mandatory to provide appropriate surgical condition. However, not only mechanical ventilation is associated with inflammatory response, but also one lung ventilation will result in detrimental effects such as ischemia and reperfusion injury, and systemic inflammatory responses.

Dexmedetomidine is an alpha-2 selective agonist. It was reported that dexmedetomidine decreased reperfusion injury, reduce the release of proinflammatory mediator and protected lungs from reperfusion injury in esophageal cancer patients who undergoing one lung ventilation from reducing oxidative stress metabolites. However, other details of protective effects is still unknown.

High mobility group box 1 (HMGB1) is an important proinflammatory factor. It was found to be related to ventilator induced lung injury in several condition. Animal studies also showed that dexmedetomidine reduces the expression of messenger ribonucleic acid in lipopolysaccharide-activated macrophage so that decrease the amount of HMGB1 release. However, clinical trials about these are still lacking.

In this study, we will investigate the protective effects of dexmedetomidine to patients undergoing video-assisted thoracoscopic surgery, especially on the specific inflammatory markers- plasma HMGB1 and other inflammatory cytokines (eg. interleukin-1. interleukin-6). This will let us to know the role of HMGB1 during one-lung ventilation injury and the effect of dexmedetomidine in regulating the release of HMGB1. This study will become a basis of further medical therapy in treating inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical classification I-II patients who receive VATS lobectomy
2. Patients with the following will be excluded:

   * suspect of infection, eg. white blood cell count> 10000 ; fever> 38.3℃
   * preoperative cardiac or renal dysfunction, eg. New York Heart Association >= II, estimated glomerular filtration rate< 60
   * predisposing liver dysfunction, eg. aspartate aminotransferase or alanine aminotransferase >100; total bilirubin> 2mg/dl; >= Child B liver cirrhosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Postoperative plasma level of HMGB1 | 2 days

SECONDARY OUTCOMES:
Postoperative complications | during hospital stay, an expected average of one week

OTHER OUTCOMES:
Postoperative pain score | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan